CLINICAL TRIAL: NCT05641935
Title: Multi-Modality Detection of RCC Recurrence Post Ablation
Brief Title: Contrast-Enhanced Ultrasound Imaging for Diagnosing Recurrent Renal Cell Carcinoma (RCC) Post Ablation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: john eisenbrey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, john eisenbrey, Associate Professor, Radiology, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22F.825; R01CA269750 (NIH); JT 24546 (Other: JeffTrial Number)
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Renal Cell Carcinoma; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic (CEUS with MRI/CT) (Experimental): Patients receive Lumason IV and undergo CEUS imaging with MRI/CT on study. Patients' electronic medical record is reviewed every 6 months throughout study.
  Interventions: Drug: Sulfur Hexafluoride Lipid Microspheres; Procedure: Contrast-Enhanced Ultrasound; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Electronic Health Record Review

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Microspheres — Given IV
  Other Names: Lumason; SF6 Lipid Microspheres; Sulfur Hexafluoride Lipid-type A Microspheres
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
  Other Names: CEUS
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging
Other: Electronic Health Record Review — Review electronic medical record

SUMMARY:
This phase II trial studies how well contrast-enhanced ultrasound (CEUS) works for diagnosing patients with renal cell cancer (RCC) that has come back (recurrent) after an ablation. Diagnostic imaging, such as CEUS, may help find and monitor long term renal cell cancer recurrence following cryo or microwave ablation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize and compare the sensitivity, specificity, positive and negative predictive value, and inter-reader agreement of 2D contrast-enhanced ultrasound (CEUS) and contrast-enhanced computed tomography (CT)/magnetic resonance imaging (MRI) for detecting recurrent or residual renal cell carcinoma (RCC) following ablation, using a combination of standard of care imaging follow-up and tissue pathology as a reference standard.

SECONDARY OBJECTIVES:

I. To evaluate the potential improvement to the qualitative assessments of 2D CEUS when fused with the patient's pre-treatment cross sectional imaging.

II. To assess the potential added value of using multi-modality volumetric CEUS for detecting RCC recurrence post ablation.

III. To explore the use of quantitative imaging parameters extracted from 2D/3D CEUS datasets to determine if this improves the overall performance of CEUS.

EXPLORATORY OBJECTIVE:

I. An advanced Doppler technique designed for detection of slower flow will also be investigated as a non-contrast based approach for detecting recurrent disease.

OUTLINE:

Patients receive Lumason intravenously (IV) and undergo CEUS imaging with MRI/CT on study. Patients' electronic medical record is reviewed every 6 months throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Previously received cryotherapy or microwave therapy of RCC
* Has available contrast enhanced (CE)-MRI or CE-CT imaging prior to ablative therapy
* Have previously had or are scheduled to have a contrast-enhanced MRI/CT for the monitoring of RCC recurrence within 4 weeks of the CEUS study
* Be at least 18 years of age
* Be medically stable
* If a female of child-bearing age, must have a negative pregnancy test
* Have signed Informed Consent to participate in the study

Exclusion Criteria:

* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable
* Patients with known sensitivities to the components of Lumason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Renal cell carcinoma recurrence | Up to 2 years
  Baseline imaging will be reviewed and compared to the contrast enhanced imaging to diagnose recurrence.

SECONDARY OUTCOMES:
Improvement of diagnostic imaging using 2D contrast-enhanced ultrasound (CEUS) with magnetic resonance/ computed tomography fusion | Up to 2 years
  Contrast-enhanced imaging on all patients will be evaluated by radiologists at each site to determine if it increases the ability to diagnose recurrence compared to standard imaging.
Measurement with multimodality 3D CEUS to improve detection of recurrence | Up to 2 years
  3D CEUS imaging will be evaluated by radiologists at each site to determine if it improved detection of recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No